CLINICAL TRIAL: NCT01251367
Title: A Phase III, Prospective, Multicentre, Open Label, Extension Study, to Assess the Long Term Safety and Efficacy of Repeated Treatment of Dysport® Intramuscular Injection in the Treatment of Lower Limb Spasticity in Adult Subjects With Spastic Hemiparesis Due to Stroke or Traumatic Brain Injury
Brief Title: Dysport® Adult Lower Limb Spasticity Follow-on Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-55-52120-142; 2009-017723-26 (EudraCT Number)
Record Dates: First submitted 2010-11-25; First posted 2010-12-01 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Post-stroke Spasticity; Spasticity Post-Traumatic Brain Injury
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport® (Experimental): Dysport® is injected into lower limbs across 4 cycles of treatment, a minimum of 12 weeks between 2 injections. Doses vary from 1000 U to 1500 U.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — I.M. (intramuscular) injection on day 1 of each treatment cycle.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this research study is to assess the long term safety of Dysport® in hemiparetic subjects with lower limb spasticity due to stroke or traumatic brain injury over repeated treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Completion of Dysport® Adult Lower Limb Spasticity Double Blind study Y-55-52120-140 (NCT01249404)

Exclusion Criteria:

* Fixed contractures in lower limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (50):
- United States (15):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Rancho Los Amigos, Downey, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - Associated Neurologist of Southern CT, PC, Fairfield, Connecticut
  - Design Neuroscience Center, Miami, Florida
  - Weill Cornell Medical College, New York, New York
  - Island Neurological Associates, Plainview, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Moss Rehab & Albert Einstein, Elkins Park, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center at Dalla, Dallas, Texas
  - University of North Texas HSC at Ben Hogan Center, Fort Worth, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Australia (6):
  - St George Hospital, Kogarah
  - Epworth Rehabilitation, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - St Vincent's Hospital, Melbourne
  - St Vincent's Hospital, Sydney
  - Westmead Hospital, Sydney
- Belgium (2):
  - Université catholique de Louvain av Hippocrate 10, Brussels
  - Clinique Universitaire, Yvoir
- Charles University in Prague, Prague, Czechia
- France (8):
  - CHU Jean MINJOZ, Besançon
  - Centre de Réadaptation de Coubert, Coubert
  - Centre Hospitalier Albert Chenevier-Hopital Henri Mondor, Créteil
  - Hopital Raymond Poincarré, Garches
  - Hôpital de L'Archet I, Nice
  - Hôpital Sébastopol, Reims
  - Hôpital Civil, Strasbourg
  - Hopital Rangueil, Toulouse
- Hungary (3):
  - National Institute for Medical Rehabilitation, Budapest
  - Uno Medical Trials, Budapest
  - Petz Aladar Country Hospital, Győr
- Azienda Ospedaliero Universitaria "Policlinico Vittorio Emanuele", Catania, Italy
- Poland (6):
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Malopolskie Centrum Medyczne, Krakow
  - Nzoz Neuro - Card, Poznan
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Portugal (3):
  - Serviço de Reabilitação, Alcabideche
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar São João, Porto
- Russia (3):
  - Medical Rehabilitation Center, Moscow
  - Scientific Research Institute of Neurology, Moscow
  - State University, Saint Petersburg
- Slovakia (2):
  - Derer's Hospital, Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Esquenazi A, Brashear A, Deltombe T, Rudzinska-Bar M, Krawczyk M, Skoromets A, O'Dell MW, Grandoulier AS, Vilain C, Picaut P, Gracies JM. The Effect of Repeated abobotulinumtoxinA (Dysport(R)) Injections on Walking Velocity in Persons with Spastic Hemiparesis Caused by Stroke or Traumatic Brain Injury. PM R. 2021 May;13(5):488-495. doi: 10.1002/pmrj.12459. Epub 2020 Sep 11. PMID 32741133
- [Derived] Esquenazi A, Stoquart G, Hedera P, Jacinto LJ, Dimanico U, Constant-Boyer F, Brashear A, Grandoulier AS, Vilain C, Picaut P, Gracies JM. Efficacy and Safety of AbobotulinumtoxinA for the Treatment of Hemiparesis in Adults with Lower Limb Spasticity Previously Treated With Other Botulinum Toxins: A Secondary Analysis of a Randomized Controlled Trial. PM R. 2020 Sep;12(9):853-860. doi: 10.1002/pmrj.12348. Epub 2020 Mar 27. PMID 32108436
- [Derived] McAllister PJ, Khatkova SE, Faux SG, Picaut P, Raymond R, Gracies JM. Effects on walking of simultaneous upper/lower limb abobotulinumtoxina injections in patients with stroke or brain injury with spastic hemiparesis. J Rehabil Med. 2019 Oct 29;51(10):813-816. doi: 10.2340/16501977-2604. PMID 31529136
- [Derived] Gracies JM, Esquenazi A, Brashear A, Banach M, Kocer S, Jech R, Khatkova S, Benetin J, Vecchio M, McAllister P, Ilkowski J, Ochudlo S, Catus F, Grandoulier AS, Vilain C, Picaut P; International AbobotulinumtoxinA Adult Lower Limb Spasticity Study Group. Efficacy and safety of abobotulinumtoxinA in spastic lower limb: Randomized trial and extension. Neurology. 2017 Nov 28;89(22):2245-2253. doi: 10.1212/WNL.0000000000004687. Epub 2017 Nov 1. PMID 29093068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed as a multicentre study and included 51 sites in Australia, Belgium, the Czech Republic, France, Hungary, Italy, Poland, Portugal, Russia, Slovakia and the United States of America that included at least one subject. The current study (Study 142) was an open label extension to the double blind Study 140 (Y-55-52120-140).
Pre-assignment Details: A total of 366 subjects completed Study 140, of which 352 subjects were enrolled in Study 142. Of these, 7 subjects entered an observational phase and never received open label treatment with Dysport® in Study 142 and the remaining 345 subjects started treatment and received at least one open label injection of Dysport® in Study 142.
Groups:
- Total Dysport®: Subjects who had completed Study 140 were offered to continue to receive open label treatment with Dysport® in Study 142 for a maximum of 4 additional treatment cycles, with a minimum interval of 12 weeks between treatment cycles. All subjects were administered an appropriate dosage of Dysport® (1500 Units [U] or 1000 U) by intramuscular (i.m.) injection in the lower limb on Day 1 of treatment Cycle 1. In all cases, the administration of the Dysport® injections was limited to a maximum dose of 1500 U every 12 weeks. Follow up visits were timed to assess the onset and progression of treatment response. From treatment Cycle 3 onwards, subjects with co-existing upper limb spasticity were able to receive concomitant injections of Dysport® into at least one upper limb muscle at a dose not exceeding 500 U. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
Period: Overall Study
Arm/Group | Total Dysport®
Started | 345
Cycle 1 | 345
Cycle 2 | 297
Cycle 3 | 224
Cycle 4 | 139
Completed | 269
Not Completed | 76
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 19
Not completed — Withdrawal by Subject | 36
Not completed — Lost to Follow-up | 5
Not completed — Subject Required Alternative Treatment | 7
Not completed — No Study Drug Available | 1
Not completed — Subject had Personal or Medical Issues | 4
Not completed — End of Study Visit Performed in Error | 1

BASELINE CHARACTERISTICS:
Population: The summary of baseline characteristics presented are from subjects completing Study 140 who were selected by the investigator for entry into Study 142 and received at least one injection of study treatment in this open label extension study.
Groups:
- Total Dysport®: Subjects who had completed Study 140 were offered to continue to receive open label treatment with Dysport® in Study 142 for a maximum of 4 additional treatment cycles, with a minimum interval of 12 weeks between treatment cycles. All subjects were administered an appropriate dosage of Dysport® (1500 U or 1000 U) by i.m. injection in the lower limb on Day 1 of treatment Cycle 1. In all cases, the administration of the Dysport® injections was limited to a maximum dose of 1500 U every 12 weeks. Follow up visits were timed to assess the onset and progression of treatment response. From treatment Cycle 3 onwards, subjects with co-existing upper limb spasticity were able to receive concomitant injections of Dysport® into at least one upper limb muscle at a dose not exceeding 500 U. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 280
  >=65 years | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 235
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34
  Not Hispanic or Latino | 311
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 21
  White | 313
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Long-Term Safety of Dysport® Through the Collection of Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were monitored from the time that the subject gave informed consent to the end of the study/early withdrawal (EOS/EW). An AE was reported as a TEAE if it was not present prior to study treatment administration in Study 140, or if it was present prior to study treatment in Study 140 but the intensity increased during the treatment phase of this study. Adverse events of special interest (AESIs) were identified as those assessed as being due to remote spread of effect of Dysport®, or any AE that was assessed as a hypersensitivity reaction. TEAEs, treatment related TEAEs, severe TEAEs, TEAEs leading to death, TEAEs leading to withdrawal, treatment emergent AESIs, and serious adverse events (SAEs) are summarised by treatment cycle.
Time Frame: Up to EOS (maximum duration of 52 weeks).
Population: Subjects who received at least one open label injection of Dysport® were included in this analysis population. The number of subjects with data available for analysis at each treatment cycle are reported.
Measure: Number; unit: participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
participants
  TEAE - Cycle 1 | 140
  TEAE - Cycle 2: number analyzed (Participants) | 297
  TEAE - Cycle 2 | 97
  TEAE - Cycle 3: number analyzed (Participants) | 224
  TEAE - Cycle 3 | 47
  TEAE - Cycle 4: number analyzed (Participants) | 139
  TEAE - Cycle 4 | 21
  Treatment Related TEAE - Cycle 1 | 43
  Treatment Related TEAE - Cycle 2: number analyzed (Participants) | 297
  Treatment Related TEAE - Cycle 2 | 23
  Treatment Related TEAE - Cycle 3: number analyzed (Participants) | 224
  Treatment Related TEAE - Cycle 3 | 7
  Treatment Related TEAE - Cycle 4: number analyzed (Participants) | 139
  Treatment Related TEAE - Cycle 4 | 5
  Severe TEAE - Cycle 1 | 13
  Severe TEAE - Cycle 2: number analyzed (Participants) | 297
  Severe TEAE - Cycle 2 | 9
  Severe TEAE - Cycle 3: number analyzed (Participants) | 224
  Severe TEAE - Cycle 3 | 4
  Severe TEAE - Cycle 4: number analyzed (Participants) | 139
  Severe TEAE - Cycle 4 | 2
  TEAE leading to death - Cycle 1 | 0
  TEAE leading to death - Cycle 2: number analyzed (Participants) | 297
  TEAE leading to death - Cycle 2 | 1
  TEAE leading to death - Cycle 3: number analyzed (Participants) | 224
  TEAE leading to death - Cycle 3 | 1
  TEAE leading to death - Cycle 4: number analyzed (Participants) | 139
  TEAE leading to death - Cycle 4 | 0
  TEAE leading to withdrawal - Cycle 1 | 8
  TEAE leading to withdrawal - Cycle 2: number analyzed (Participants) | 297
  TEAE leading to withdrawal - Cycle 2 | 10
  TEAE leading to withdrawal - Cycle 3: number analyzed (Participants) | 224
  TEAE leading to withdrawal - Cycle 3 | 1
  TEAE leading to withdrawal - Cycle 4: number analyzed (Participants) | 139
  TEAE leading to withdrawal - Cycle 4 | 0
  AESI - Cycle 1 | 31
  AESI - Cycle 2: number analyzed (Participants) | 297
  AESI - Cycle 2 | 24
  AESI - Cycle 3: number analyzed (Participants) | 224
  AESI - Cycle 3 | 10
  AESI - Cycle 4: number analyzed (Participants) | 139
  AESI - Cycle 4 | 5
  SAE - Cycle 1 | 23
  SAE - Cycle 2: number analyzed (Participants) | 297
  SAE - Cycle 2 | 14
  SAE - Cycle 3: number analyzed (Participants) | 224
  SAE - Cycle 3 | 7
  SAE - Cycle 4: number analyzed (Participants) | 139
  SAE - Cycle 4 | 2

2. Primary Outcome: Mean Change From Baseline to Week 4 in Systolic and Diastolic Blood Pressure (BP)
Description: Systolic and diastolic BP were recorded at baseline and at each subsequent study visit. BP was measured with the subject in a sitting position after resting for 3 minutes. Mean change in BP from baseline at Week 4 is reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: Millimetres Mercury (mmHg)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Millimetres Mercury (mmHg)
  Systolic BP - Cycle 1: number analyzed (Participants) | 331
  Systolic BP - Cycle 1 | -0.7 [-67 to 37]
  Systolic BP - Cycle 2: number analyzed (Participants) | 281
  Systolic BP - Cycle 2 | -1.9 [-69 to 37]
  Systolic BP - Cycle 3: number analyzed (Participants) | 200
  Systolic BP - Cycle 3 | -2.4 [-58 to 79]
  Systolic BP - Cycle 4: number analyzed (Participants) | 92
  Systolic BP - Cycle 4 | -5.1 [-73 to 25]
  Diastolic BP - Cycle 1: number analyzed (Participants) | 331
  Diastolic BP - Cycle 1 | 0.3 [-34 to 37]
  Diastolic BP - Cycle 2: number analyzed (Participants) | 281
  Diastolic BP - Cycle 2 | -0.2 [-38 to 30]
  Diastolic BP - Cycle 3: number analyzed (Participants) | 200
  Diastolic BP - Cycle 3 | -0.3 [-32 to 28]
  Diastolic BP - Cycle 4: number analyzed (Participants) | 92
  Diastolic BP - Cycle 4 | -1.1 [-35 to 32]

3. Primary Outcome: Mean Change From Baseline to Week 4 in Heart Rate (HR)
Description: HR was recorded at baseline and at each subsequent study visit. HR was measured with the subject in a sitting position after resting for 3 minutes. Mean change in HR from baseline at Week 4 is reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: Beats per minute (bpm)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Beats per minute (bpm)
  Cycle 1: number analyzed (Participants) | 331
  Cycle 1 | 3.7 [-28 to 39]
  Cycle 2: number analyzed (Participants) | 281
  Cycle 2 | 4.9 [-27 to 41]
  Cycle 3: number analyzed (Participants) | 200
  Cycle 3 | 3.9 [-25 to 52]
  Cycle 4: number analyzed (Participants) | 92
  Cycle 4 | 4.5 [-16 to 33]

4. Primary Outcome: Mean Change From Baseline to Week 4 in Red Blood Cell (RBC) Count
Description: Blood samples for RBC count were taken at baseline, at Week 4, and at EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: Tera cells/Litre (L)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Tera cells/Litre (L)
  Cycle 1: number analyzed (Participants) | 305
  Cycle 1 | 0.049 [-0.51 to 0.66]
  Cycle 2: number analyzed (Participants) | 260
  Cycle 2 | 0.074 [-0.59 to 0.68]
  Cycle 3: number analyzed (Participants) | 180
  Cycle 3 | 0.046 [-0.59 to 0.66]
  Cycle 4: number analyzed (Participants) | 78
  Cycle 4 | 0.028 [-1.24 to 0.61]

5. Primary Outcome: Mean Change From Baseline to Week 4 in Haemoglobin and Mean Corpuscular Haemoglobin Concentration (MCHC)
Description: Blood samples for haemoglobin and MCHC were taken at baseline, at Week 4, and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: grams (g)/L
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
grams (g)/L
  Haemoglobin - Cycle 1: number analyzed (Participants) | 305
  Haemoglobin - Cycle 1 | 1.2 [-17 to 32]
  Haemoglobin - Cycle 2: number analyzed (Participants) | 260
  Haemoglobin - Cycle 2 | 1.5 [-46 to 25]
  Haemoglobin - Cycle 3: number analyzed (Participants) | 180
  Haemoglobin - Cycle 3 | 1.5 [-22 to 26]
  Haemoglobin - Cycle 4: number analyzed (Participants) | 78
  Haemoglobin - Cycle 4 | 1.2 [-39 to 17]
  MCHC - Cycle 1: number analyzed (Participants) | 305
  MCHC - Cycle 1 | 1.9 [-29 to 34]
  MCHC - Cycle 2: number analyzed (Participants) | 260
  MCHC - Cycle 2 | 1.3 [-33 to 41]
  MCHC - Cycle 3: number analyzed (Participants) | 180
  MCHC - Cycle 3 | 3.4 [-23 to 33]
  MCHC - Cycle 4: number analyzed (Participants) | 78
  MCHC - Cycle 4 | 8.9 [-14 to 37]

6. Primary Outcome: Mean Change From Baseline to Week 4 in Haematocrit
Description: Blood samples for haematocrit were taken at baseline, at Week 4, and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of RBC in blood
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
percentage of RBC in blood
  Cycle 1: number analyzed (Participants) | 305
  Cycle 1 | 0.001 [-0.057 to 0.081]
  Cycle 2: number analyzed (Participants) | 260
  Cycle 2 | 0.003 [-0.107 to 0.098]
  Cycle 3: number analyzed (Participants) | 180
  Cycle 3 | -0.001 [-0.066 to 0.086]
  Cycle 4: number analyzed (Participants) | 78
  Cycle 4 | -0.009 [-0.12 to 0.047]

7. Primary Outcome: Mean Change From Baseline to Week 4 in Mean Corpuscular Haemoglobin (MCH)
Description: Blood samples for MCH were taken at baseline, at Week 4, and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: picograms (pg)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
picograms (pg)
  Cycle 1: number analyzed (Participants) | 305
  Cycle 1 | -0.06 [-4.7 to 6.3]
  Cycle 2: number analyzed (Participants) | 260
  Cycle 2 | -0.17 [-9.3 to 4.6]
  Cycle 3: number analyzed (Participants) | 180
  Cycle 3 | 0.00 [-2.8 to 5.3]
  Cycle 4: number analyzed (Participants) | 78
  Cycle 4 | 0.05 [-1.8 to 2]

8. Primary Outcome: Mean Change From Baseline to Week 4 in Mean Corpuscular Volume (MCV)
Description: Blood samples for MCV were taken at baseline, at Week 4, and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: Femtolitres (fL)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Femtolitres (fL)
  Cycle 1: number analyzed (Participants) | 305
  Cycle 1 | -0.74 [-10.3 to 14.8]
  Cycle 2: number analyzed (Participants) | 260
  Cycle 2 | -0.9 [-21.2 to 12.5]
  Cycle 3: number analyzed (Participants) | 180
  Cycle 3 | -1.02 [-8.5 to 13.7]
  Cycle 4: number analyzed (Participants) | 78
  Cycle 4 | -2.44 [-9.1 to 3.7]

9. Primary Outcome: Mean Change From Baseline to Week 4 in White Blood Cell (WBC) Count, Neutrophils, Lymphocytes and Platelets
Description: Blood samples for WBC count with differentials (neutrophils, lymphocytes) and platelet count were taken at baseline, at Week 4, and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: Giga cells/L
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Giga cells/L
  WBC count - Cycle 1: number analyzed (Participants) | 305
  WBC count - Cycle 1 | -0.21 [-8.7 to 5.3]
  WBC count - Cycle 2: number analyzed (Participants) | 260
  WBC count - Cycle 2 | -0.32 [-5.7 to 4.9]
  WBC count - Cycle 3: number analyzed (Participants) | 180
  WBC count - Cycle 3 | -0.26 [-5.2 to 5.1]
  WBC count - Cycle 4: number analyzed (Participants) | 78
  WBC count - Cycle 4 | -0.02 [-4.3 to 5.2]
  Neutrophils - Cycle 1: number analyzed (Participants) | 304
  Neutrophils - Cycle 1 | -0.17 [-7.5 to 4.5]
  Neutrophils - Cycle 2: number analyzed (Participants) | 259
  Neutrophils - Cycle 2 | -0.27 [-5.3 to 4.2]
  Neutrophils - Cycle 3: number analyzed (Participants) | 179
  Neutrophils - Cycle 3 | -0.28 [-5.6 to 4.8]
  Neutrophils - Cycle 4: number analyzed (Participants) | 78
  Neutrophils - Cycle 4 | -0.06 [-4.4 to 5.5]
  Lymphocytes - Cycle 1: number analyzed (Participants) | 303
  Lymphocytes - Cycle 1 | -0.05 [-1.3 to 1.4]
  Lymphocytes - Cycle 2: number analyzed (Participants) | 258
  Lymphocytes - Cycle 2 | -0.05 [-1.3 to 1.4]
  Lymphocytes - Cycle 3: number analyzed (Participants) | 179
  Lymphocytes - Cycle 3 | 0.03 [-1.2 to 2.5]
  Lymphocytes - Cycle 4: number analyzed (Participants) | 78
  Lymphocytes - Cycle 4 | -0.01 [-0.9 to 2]
  Platelets - Cycle 1: number analyzed (Participants) | 300
  Platelets - Cycle 1 | -0.1 [-193 to 192]
  Platelets - Cycle 2: number analyzed (Participants) | 257
  Platelets - Cycle 2 | 0.0 [-133 to 276]
  Platelets - Cycle 3: number analyzed (Participants) | 178
  Platelets - Cycle 3 | 0.1 [-139 to 152]
  Platelets - Cycle 4: number analyzed (Participants) | 77
  Platelets - Cycle 4 | 4.6 [-67 to 167]

10. Primary Outcome: Mean Change From Baseline to Week 4 in Alkaline Phosphatase (ALP), Gamma Glutamyl Transferase (GGT), Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase (SGPT)
Description: Blood samples were taken at baseline, at Week 4, and at the EOS/EW for analysis of the following clinical chemistry parameters: ALP, GGT, SGOT and SGPT. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
IU/L
  ALP - Cycle 1: number analyzed (Participants) | 319
  ALP - Cycle 1 | -1.2 [-60 to 110]
  ALP - Cycle 2: number analyzed (Participants) | 268
  ALP - Cycle 2 | -2.9 [-141 to 57]
  ALP - Cycle 3: number analyzed (Participants) | 188
  ALP - Cycle 3 | -5.2 [-238 to 33]
  ALP - Cycle 4: number analyzed (Participants) | 85
  ALP - Cycle 4 | -3.2 [-45 to 39]
  SGOT - Cycle 1: number analyzed (Participants) | 319
  SGOT - Cycle 1 | 2.7 [-47 to 35]
  SGOT - Cycle 2: number analyzed (Participants) | 268
  SGOT - Cycle 2 | 3 [-27 to 144]
  SGOT - Cycle 3: number analyzed (Participants) | 188
  SGOT - Cycle 3 | 1.3 [-109 to 34]
  SGOT - Cycle 4: number analyzed (Participants) | 85
  SGOT - Cycle 4 | 1.8 [-12 to 19]
  SGPT - Cycle 1: number analyzed (Participants) | 319
  SGPT - Cycle 1 | 1.2 [-60 to 45]
  SGPT - Cycle 2: number analyzed (Participants) | 268
  SGPT - Cycle 2 | 2.4 [-53 to 302]
  SGPT - Cycle 3: number analyzed (Participants) | 188
  SGPT - Cycle 3 | 1.7 [-444 to 69]
  SGPT - Cycle 4: number analyzed (Participants) | 85
  SGPT - Cycle 4 | 0.8 [-28 to 25]
  GGT - Cycle 1: number analyzed (Participants) | 320
  GGT - Cycle 1 | 1 [-122 to 614]
  GGT - Cycle 2: number analyzed (Participants) | 268
  GGT - Cycle 2 | -1.9 [-145 to 121]
  GGT - Cycle 3: number analyzed (Participants) | 188
  GGT - Cycle 3 | -3 [-254 to 107]
  GGT - Cycle 4: number analyzed (Participants) | 85
  GGT - Cycle 4 | -0.4 [-61 to 70]

11. Primary Outcome: Mean Change From Baseline to Week 4 in Total Bilirubin and Creatinine
Description: Blood samples for clinical chemistry analysis of total bilirubin and creatinine were taken at baseline, at Week 4, and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: Micromole/L (μmol/L)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Micromole/L (μmol/L)
  Total bilirubin - Cycle 1: number analyzed (Participants) | 319
  Total bilirubin - Cycle 1 | 0.13 [-13.7 to 12.8]
  Total bilirubin - Cycle 2: number analyzed (Participants) | 268
  Total bilirubin - Cycle 2 | 0.14 [-10.6 to 15.2]
  Total bilirubin - Cycle 3: number analyzed (Participants) | 188
  Total bilirubin - Cycle 3 | 0.03 [-10.4 to 7]
  Total bilirubin - Cycle 4: number analyzed (Participants) | 85
  Total bilirubin - Cycle 4 | -0.05 [-9.1 to 16.1]
  Creatinine - Cycle 1: number analyzed (Participants) | 320
  Creatinine - Cycle 1 | -2 [-36 to 27]
  Creatinine - Cycle 2: number analyzed (Participants) | 268
  Creatinine - Cycle 2 | -5.3 [-36 to 35]
  Creatinine - Cycle 3: number analyzed (Participants) | 188
  Creatinine - Cycle 3 | -7.9 [-53 to 35]
  Creatinine - Cycle 4: number analyzed (Participants) | 85
  Creatinine - Cycle 4 | -14.2 [-62 to 9]

12. Primary Outcome: Mean Change From Baseline to Week 4 in Blood Urea Nitrogen (BUN) and Fasting Blood Glucose
Description: Blood samples for analysis of BUN and fasting blood glucose levels were taken at baseline, at Week 4 and at the EOS/EW. Outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Full Range); unit: millimole/L (mmol/L)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
millimole/L (mmol/L)
  BUN - Cycle 1: number analyzed (Participants) | 320
  BUN - Cycle 1 | 0.14 [-3.93 to 5]
  BUN - Cycle 2: number analyzed (Participants) | 268
  BUN - Cycle 2 | -0.05 [-3.57 to 5.72]
  BUN - Cycle 3: number analyzed (Participants) | 188
  BUN - Cycle 3 | -0.19 [-11.06 to 4.29]
  BUN - Cycle 4: number analyzed (Participants) | 85
  BUN - Cycle 4 | -0.37 [-4.64 to 3.57]
  Fasting blood glucose - Cycle 1: number analyzed (Participants) | 169
  Fasting blood glucose - Cycle 1 | -0.046 [-6.16 to 6.38]
  Fasting blood glucose - Cycle 2: number analyzed (Participants) | 143
  Fasting blood glucose - Cycle 2 | 0.009 [-4.17 to 9.44]
  Fasting blood glucose - Cycle 3: number analyzed (Participants) | 101
  Fasting blood glucose - Cycle 3 | 0.015 [-5.66 to 7]
  Fasting blood glucose - Cycle 4: number analyzed (Participants) | 55
  Fasting blood glucose - Cycle 4 | 0.231 [-3.44 to 8.61]

13. Primary Outcome: Presence of Botulinum Toxin Type A (BTX-A) Neutralising Putative Antibodies (NAbs) Following Injection of Dysport®
Description: Blood samples were collected at baseline, Week 4 and at EOS/EW to test for the presence of BTX-A antibodies. The number of subjects who were either NAb positive at baseline or negative at baseline but then positive following injection of Dysport® were reported.
Time Frame: At Week 4
Population: Subjects who received at least one open label injection of Dysport® were included in this analysis population. In addition, the antibody analysis included subjects who had an antibody assessment at baseline and at a post baseline visit (n=343).
Measure: Count of Participants; unit: Participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Participants
  Positive at baseline: number analyzed (Participants) | 343
  Positive at baseline | 3
  Negative at baseline & positive post baseline: number analyzed (Participants) | 343
  Negative at baseline & positive post baseline | 0

14. Primary Outcome: Mean Change From Baseline to Week 4 in 12-Lead Electrocardiogram (ECG)
Description: 12-lead ECG tracing was performed at baseline, at Week 4 of each cycle and at EOS/EW. The 12-lead ECG recordings were performed at a paper speed of 25 millimetres/second (mm/s), recorded with the subject in a supine position after 5 minutes rest. The ECG parameters; QT Duration, QT interval corrected with Fridericia's method (QTcF), QT interval corrected with Bazett's method (QTcB), QRS duration and PR duration were recorded and outcome measure is reported per cycle as change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: Subjects who received at least one open label injection of Dysport® were included in this analysis population.
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 324
Milliseconds (ms)
  QT Duration - Cycle 1: number analyzed (Participants) | 301
  QT Duration - Cycle 1 | -10.1 (24.9)
  QT Duration - Cycle 2: number analyzed (Participants) | 260
  QT Duration - Cycle 2 | -12.2 (22.9)
  QT Duration - Cycle 3: number analyzed (Participants) | 181
  QT Duration - Cycle 3 | -13.6 (26.5)
  QT Duration - Cycle 4: number analyzed (Participants) | 83
  QT Duration - Cycle 4 | -16.5 (23.5)
  QTcF - Cycle 1: number analyzed (Participants) | 301
  QTcF - Cycle 1 | -0.6 (16.9)
  QTcF - Cycle 2: number analyzed (Participants) | 260
  QTcF - Cycle 2 | -1.9 (14.8)
  QTcF - Cycle 3: number analyzed (Participants) | 181
  QTcF - Cycle 3 | -3.8 (16.2)
  QTcF - Cycle 4: number analyzed (Participants) | 83
  QTcF - Cycle 4 | -1.8 (16.1)
  QTcB - Cycle 1: number analyzed (Participants) | 301
  QTcB - Cycle 1 | 4.5 (20.2)
  QTcB - Cycle 2: number analyzed (Participants) | 260
  QTcB - Cycle 2 | 3.5 (18.4)
  QTcB - Cycle 3: number analyzed (Participants) | 181
  QTcB - Cycle 3 | 1.5 (19.5)
  QTcB - Cycle 4: number analyzed (Participants) | 83
  QTcB - Cycle 4 | 6.1 (21.3)
  QRS Duration - Cycle 1: number analyzed (Participants) | 301
  QRS Duration - Cycle 1 | -0.6 (6.3)
  QRS Duration - Cycle 2: number analyzed (Participants) | 260
  QRS Duration - Cycle 2 | -0.7 (5.8)
  QRS Duration - Cycle 3: number analyzed (Participants) | 181
  QRS Duration - Cycle 3 | -0.8 (6.2)
  QRS Duration - Cycle 4: number analyzed (Participants) | 83
  QRS Duration - Cycle 4 | -0.9 (6.7)
  PR Duration - Cycle 1: number analyzed (Participants) | 300
  PR Duration - Cycle 1 | -2.2 (14.5)
  PR Duration - Cycle 2: number analyzed (Participants) | 259
  PR Duration - Cycle 2 | -1.7 (15.2)
  PR Duration - Cycle 3: number analyzed (Participants) | 181
  PR Duration - Cycle 3 | -0.5 (14.4)
  PR Duration - Cycle 4: number analyzed (Participants) | 83
  PR Duration - Cycle 4 | -0.6 (13.4)

15. Secondary Outcome: Mean Change From Baseline to Week 4 in the Modified Ashworth Scale (MAS) Score Measured in the Gastrocnemius-soleus Complex (GSC) (Knee Extended)
Description: Muscle tone in the treated limb was assessed by MAS in the GSC (with the knee extended) at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM)), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. Outcome measure is reported per cycle as mean change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Cycle 1: number analyzed (Participants) | 341
  Cycle 1 | -0.8 (0.9)
  Cycle 2: number analyzed (Participants) | 290
  Cycle 2 | -0.9 (1)
  Cycle 3: number analyzed (Participants) | 218
  Cycle 3 | -1 (1)
  Cycle 4: number analyzed (Participants) | 135
  Cycle 4 | -1 (0.9)

16. Secondary Outcome: Mean Change From Baseline to Week 4 in the MAS Measured in the Soleus Muscle (Knee Flexed)
Description: Muscle tone in the treated limb was assessed by MAS in the soleus muscle (with the knee flexed) at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. Outcome measure is reported per cycle as mean change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Cycle 1: number analyzed (Participants) | 340
  Cycle 1 | -1 (1.2)
  Cycle 2: number analyzed (Participants) | 290
  Cycle 2 | -1.1 (1)
  Cycle 3: number analyzed (Participants) | 218
  Cycle 3 | -1.2 (1)
  Cycle 4: number analyzed (Participants) | 135
  Cycle 4 | -1.1 (1.1)

17. Secondary Outcome: Percentage of Subjects With At Least a 1 or 2 Grade Reduction in the MAS Measured in the GSC (Knee Extended) at Week 4
Description: Muscle tone in the treated limb was assessed by MAS in the GSC (with the knee extended) at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. Outcome measure is reported per cycle as the percentage of subjects with at least a 1 grade reduction or 2 grades reduction in MAS score at Week 4.
Time Frame: Week 4 of each cycle
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
percentage of participants
  At least 1 grade reduction - Cycle 1 | 56.2
  At least 1 grade reduction - Cycle 2: number analyzed (Participants) | 297
  At least 1 grade reduction - Cycle 2 | 57.6
  At least 1 grade reduction - Cycle 3: number analyzed (Participants) | 224
  At least 1 grade reduction - Cycle 3 | 60.7
  At least 1 grade reduction - Cycle 4: number analyzed (Participants) | 139
  At least 1 grade reduction - Cycle 4 | 66.9
  At least 2 grades reduction - Cycle 1 | 18.3
  At least 2 grades reduction - Cycle 2: number analyzed (Participants) | 297
  At least 2 grades reduction - Cycle 2 | 23.2
  At least 2 grades reduction - Cycle 3: number analyzed (Participants) | 224
  At least 2 grades reduction - Cycle 3 | 23.2
  At least 2 grades reduction - Cycle 4: number analyzed (Participants) | 139
  At least 2 grades reduction - Cycle 4 | 22.3

18. Secondary Outcome: Percentage of Subjects With At Least a 1 or 2 Grade Reduction in the MAS Measured in the Soleus Muscle (Knee Flexed) at Week 4
Description: Muscle tone in the treated limb was assessed by MAS in the soleus muscle (with the knee flexed) at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. The MAS consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM), 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension), and can be applied to muscles of both the upper and lower limbs. Outcome measure is reported per cycle as the percentage of subjects with at least a 1 grade reduction or 2 grades reduction in MAS score at Week 4.
Time Frame: Week 4 of each cycle
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
percentage of participants
  At least 1 grade reduction - Cycle 1 | 61.4
  At least 1 grade reduction - Cycle 2: number analyzed (Participants) | 297
  At least 1 grade reduction - Cycle 2 | 68.4
  At least 1 grade reduction - Cycle 3: number analyzed (Participants) | 224
  At least 1 grade reduction - Cycle 3 | 72.3
  At least 1 grade reduction - Cycle 4: number analyzed (Participants) | 139
  At least 1 grade reduction - Cycle 4 | 71.9
  At least 2 grades reduction - Cycle 1 | 28.4
  At least 2 grades reduction - Cycle 2: number analyzed (Participants) | 297
  At least 2 grades reduction - Cycle 2 | 30.6
  At least 2 grades reduction - Cycle 3: number analyzed (Participants) | 224
  At least 2 grades reduction - Cycle 3 | 30.4
  At least 2 grades reduction - Cycle 4: number analyzed (Participants) | 139
  At least 2 grades reduction - Cycle 4 | 28.8

19. Secondary Outcome: Physician's Global Assessment (PGA) of Treatment Response at Week 4
Description: An assessment of overall treatment response was conducted by the investigator at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. The investigator rated the response to treatment in the subject's lower limb after injection of Dysport® relative to the status at the baseline. Answers were made on a nine-point rating scale: -4=markedly worse, -3=much worse, -2=worse, -1=slightly worse, 0=no change, +1=slightly improved, +2=improved, +3=much improved, +4=markedly improved. The mean PGA scores per cycle at Week 4 were reported.
Time Frame: Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Cycle 1: number analyzed (Participants) | 340
  Cycle 1 | 1.4 (1.1)
  Cycle 2: number analyzed (Participants) | 288
  Cycle 2 | 1.6 (1)
  Cycle 3: number analyzed (Participants) | 216
  Cycle 3 | 1.8 (1)
  Cycle 4: number analyzed (Participants) | 134
  Cycle 4 | 1.9 (1)

20. Secondary Outcome: Percentage of Subjects With a Score of at Least +1 on the PGA Scale at Week 4
Description: An assessment of overall treatment response was conducted by the investigator at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. The investigator rated the response to treatment in the subject's lower limb after injection of Dysport® relative to the status at the baseline. Answers were made on a nine point rating scale: -4=markedly worse, -3=much worse, -2=worse, -1=slightly worse, 0=no change, +1=slightly improved, +2=improved, +3=much improved, +4=markedly improved. The percentage of responders with a PGA score of +1 or greater are reported at Week 4.
Time Frame: Week 4 of each cycle
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
percentage of participants
  Cycle 1 | 83.8
  Cycle 2: number analyzed (Participants) | 297
  Cycle 2 | 86.2
  Cycle 3: number analyzed (Participants) | 224
  Cycle 3 | 89.3
  Cycle 4: number analyzed (Participants) | 139
  Cycle 4 | 89.9

21. Secondary Outcome: Mean Change From Baseline to Week 4 in the Range of Active Ankle Dorsiflexion Both With the Knee Flexed and With the Knee Extended
Description: Range of active dorsiflexion of the ankle joint of the treated limb, measured using a goniometre, both with the knee flexed (90°) and extended, was used to assess treatment response. The measurements were obtained at the end of baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. Outcome measure is reported per cycle as mean change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Degrees
  Knee Extended - Cycle 1: number analyzed (Participants) | 340
  Knee Extended - Cycle 1 | 4.1 (10.6)
  Knee Extended - Cycle 2: number analyzed (Participants) | 290
  Knee Extended - Cycle 2 | 4.4 (10.6)
  Knee Extended - Cycle 3: number analyzed (Participants) | 218
  Knee Extended - Cycle 3 | 6 (11.4)
  Knee Extended - Cycle 4: number analyzed (Participants) | 135
  Knee Extended - Cycle 4 | 6.5 (10.9)
  Knee Flexed - Cycle 1: number analyzed (Participants) | 341
  Knee Flexed - Cycle 1 | 4.1 (10.7)
  Knee Flexed - Cycle 2: number analyzed (Participants) | 290
  Knee Flexed - Cycle 2 | 5 (10.3)
  Knee Flexed - Cycle 3: number analyzed (Participants) | 218
  Knee Flexed - Cycle 3 | 5.2 (10.9)
  Knee Flexed - Cycle 4: number analyzed (Participants) | 135
  Knee Flexed - Cycle 4 | 3.8 (9.8)

22. Secondary Outcome: Mean Change From Baseline to Week 4 in Lower Limb Pain
Description: The intensity of lower limb pain in the treated limb was evaluated by the subject using the Scale of Pain Intensity (SPIN) which provided a pictorial representation of pain in a 6-point graphic scale with the degree of red shading inside a circle representing the intensity of pain. The bottom and top of the scale are anchored by two extremes: 'no pain' (circle with no red shading and scored as 0) and 'pain as bad as it could be' (circle completely red and scored as 5), marked with either verbal or visual cues. The intervening points are represented by red circles increasing proportionally in size. The subject marks the circle that best indicates their pain intensity. The SPIN assessments were obtained at baseline, Weeks 4 and 12 after each Dysport® injection, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at the EOS/EW. The mean changes from baseline in subjects with a baseline SPIN Score >0 at Week 4 was reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Cycle 1: number analyzed (Participants) | 189
  Cycle 1 | -0.7 (1.2)
  Cycle 2: number analyzed (Participants) | 160
  Cycle 2 | -0.8 (1.2)
  Cycle 3: number analyzed (Participants) | 118
  Cycle 3 | -0.9 (1.2)
  Cycle 4: number analyzed (Participants) | 75
  Cycle 4 | -0.9 (1.2)

23. Secondary Outcome: Mean Change From Baseline to Week 4 in Short Form (36) Health Survey (SF-36) Quality of Life (QoL)
Description: Subjects were asked to complete the SF-36 health surveys prior to the study treatment at baseline, at Week 4 and at the EOS/EW visit. The SF-36 is a generic non preference based health status measure. This instrument assessed subject health across 8 variable dimensions, which are specific health domains such as physical functioning, social functioning and vitality. Each variable item score is coded and turned into a 0-100 scale where 0 indicates the worst and 100 indicates the best possible health state for both the Physical Component Summary (PCS) and Mental Component Summary (MCS) of the questionnaire. The mean change in the PCS and MCS from baseline to Week 4 are reported.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  PCS - Cycle 1: number analyzed (Participants) | 330
  PCS - Cycle 1 | 1.05 (7.5)
  PCS - Cycle 2: number analyzed (Participants) | 287
  PCS - Cycle 2 | 1.43 (7.67)
  PCS - Cycle 3: number analyzed (Participants) | 213
  PCS - Cycle 3 | 1.85 (7.01)
  PCS - Cycle 4: number analyzed (Participants) | 134
  PCS - Cycle 4 | 2.8 (6.65)
  MCS - Cycle 1: number analyzed (Participants) | 330
  MCS - Cycle 1 | -1.13 (11.27)
  MCS - Cycle 2: number analyzed (Participants) | 287
  MCS - Cycle 2 | -0.82 (12.7)
  MCS - Cycle 3: number analyzed (Participants) | 213
  MCS - Cycle 3 | 0.56 (12.24)
  MCS - Cycle 4: number analyzed (Participants) | 134
  MCS - Cycle 4 | 0.14 (13.23)

24. Secondary Outcome: Mean Change From Baseline in European Quality of Life - 5 Dimensions, 5 Level (EQ-5D-5L) QoL
Description: Subjects were asked to complete the EQ-5D-5L QoL questionnaire prior to the study treatment at baseline, at Week 4 and at EOS/EW visit. The EQ-5D-5L index is a generic preference based measure of health related QoL producing utility scores that represent subject preferences for particular health states. This instrument rated subject health state looking at 5 specific dimensions such as mobility, self-care, usual activity, pain/discomfort and anxiety/ depression and scored their general health state. Each dimension has 5 levels of severity: no problems, slight problems, moderate problems, severe problems and extreme problems, rated from 1 to 5 (best to worst). In addition, a visual analogue scale (VAS) ranging from 0 to 100 was also included for the patients to summarize their overall health status, where 0 is the worst and 100 the best possible health state. The mean change in pain and discomfort and VAS scores from baseline to Week 4 are reported.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Pain/discomfort - Cycle 1: number analyzed (Participants) | 337
  Pain/discomfort - Cycle 1 | -0.1 (1.0)
  Pain/discomfort - Cycle 2: number analyzed (Participants) | 288
  Pain/discomfort - Cycle 2 | -0.2 (1.0)
  Pain/discomfort - Cycle 3: number analyzed (Participants) | 215
  Pain/discomfort - Cycle 3 | -0.2 (1.0)
  Pain/discomfort - Cycle 4: number analyzed (Participants) | 133
  Pain/discomfort - Cycle 4 | -0.4 (1.2)
  VAS - Cycle 1: number analyzed (Participants) | 336
  VAS - Cycle 1 | 2.8 (18.3)
  VAS - Cycle 2: number analyzed (Participants) | 286
  VAS - Cycle 2 | 3.8 (17.7)
  VAS - Cycle 3: number analyzed (Participants) | 215
  VAS - Cycle 3 | 4.4 (19.9)
  VAS - Cycle 4: number analyzed (Participants) | 133
  VAS - Cycle 4 | 5.5 (21.0)

25. Secondary Outcome: Mean Change From Baseline to Week 4 in Walking Speed (WS)
Description: All WS tests were conducted without walking aids over a distance of 10 metres at both a comfortable WS and at maximal WS. Evaluations of WS were made barefoot and with shoes on, at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. Outcome measure is reported per cycle as mean change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: metres/second (m/s)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
metres/second (m/s)
  Comfortable WS, barefoot - Cycle 1: number analyzed (Participants) | 335
  Comfortable WS, barefoot - Cycle 1 | 0.07 (0.12)
  Comfortable WS, barefoot - Cycle 2: number analyzed (Participants) | 285
  Comfortable WS, barefoot - Cycle 2 | 0.08 (0.13)
  Comfortable WS, barefoot - Cycle 3: number analyzed (Participants) | 215
  Comfortable WS, barefoot - Cycle 3 | 0.08 (0.13)
  Comfortable WS, barefoot - Cycle 4: number analyzed (Participants) | 134
  Comfortable WS, barefoot - Cycle 4 | 0.09 (0.14)
  Comfortable WS, with shoes - Cycle 1: number analyzed (Participants) | 336
  Comfortable WS, with shoes - Cycle 1 | 0.06 (0.13)
  Comfortable WS, with shoes - Cycle 2: number analyzed (Participants) | 289
  Comfortable WS, with shoes - Cycle 2 | 0.07 (0.14)
  Comfortable WS, with shoes - Cycle 3: number analyzed (Participants) | 217
  Comfortable WS, with shoes - Cycle 3 | 0.08 (0.13)
  Comfortable WS, with shoes - Cycle 4: number analyzed (Participants) | 134
  Comfortable WS, with shoes - Cycle 4 | 0.08 (0.14)
  Maximal WS, barefoot - Cycle 1: number analyzed (Participants) | 336
  Maximal WS, barefoot - Cycle 1 | 0.07 (0.16)
  Maximal WS, barefoot - Cycle 2: number analyzed (Participants) | 286
  Maximal WS, barefoot - Cycle 2 | 0.08 (0.18)
  Maximal WS, barefoot - Cycle 3: number analyzed (Participants) | 215
  Maximal WS, barefoot - Cycle 3 | 0.09 (0.18)
  Maximal WS, barefoot - Cycle 4: number analyzed (Participants) | 134
  Maximal WS, barefoot - Cycle 4 | 0.1 (0.18)
  Maximal WS, with shoes - Cycle 1: number analyzed (Participants) | 335
  Maximal WS, with shoes - Cycle 1 | 0.07 (0.17)
  Maximal WS, with shoes - Cycle 2: number analyzed (Participants) | 286
  Maximal WS, with shoes - Cycle 2 | 0.09 (0.19)
  Maximal WS, with shoes - Cycle 3: number analyzed (Participants) | 217
  Maximal WS, with shoes - Cycle 3 | 0.09 (0.19)
  Maximal WS, with shoes - Cycle 4: number analyzed (Participants) | 134
  Maximal WS, with shoes - Cycle 4 | 0.1 (0.21)

26. Secondary Outcome: Mean Change From Baseline to Week 4 in Step Length
Description: All WS tests were conducted without walking aids over a distance of 10 metres at both a comfortable WS and at maximal WS. Evaluations of step length were made barefoot and with shoes on, at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. Outcome measure is reported per cycle as mean change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/step
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
m/step
  Comfortable WS, barefoot - Cycle 1: number analyzed (Participants) | 335
  Comfortable WS, barefoot - Cycle 1 | 0.03 (0.06)
  Comfortable WS, barefoot - Cycle 2: number analyzed (Participants) | 285
  Comfortable WS, barefoot - Cycle 2 | 0.03 (0.09)
  Comfortable WS, barefoot - Cycle 3: number analyzed (Participants) | 215
  Comfortable WS, barefoot - Cycle 3 | 0.03 (0.08)
  Comfortable WS, barefoot - Cycle 4: number analyzed (Participants) | 134
  Comfortable WS, barefoot - Cycle 4 | 0.05 (0.09)
  Comfortable WS, with shoes - Cycle 1: number analyzed (Participants) | 336
  Comfortable WS, with shoes - Cycle 1 | 0.03 (0.07)
  Comfortable WS, with shoes - Cycle 2: number analyzed (Participants) | 289
  Comfortable WS, with shoes - Cycle 2 | 0.03 (0.08)
  Comfortable WS, with shoes - Cycle 3: number analyzed (Participants) | 217
  Comfortable WS, with shoes - Cycle 3 | 0.03 (0.08)
  Comfortable WS, with shoes - Cycle 4: number analyzed (Participants) | 134
  Comfortable WS, with shoes - Cycle 4 | 0.04 (0.09)
  Maximal WS, barefoot - Cycle 1: number analyzed (Participants) | 336
  Maximal WS, barefoot - Cycle 1 | 0.03 (0.08)
  Maximal WS, barefoot - Cycle 2: number analyzed (Participants) | 286
  Maximal WS, barefoot - Cycle 2 | 0.03 (0.09)
  Maximal WS, barefoot - Cycle 3: number analyzed (Participants) | 215
  Maximal WS, barefoot - Cycle 3 | 0.03 (0.09)
  Maximal WS, barefoot - Cycle 4: number analyzed (Participants) | 134
  Maximal WS, barefoot - Cycle 4 | 0.04 (0.09)
  Maximal WS, with shoes - Cycle 1: number analyzed (Participants) | 335
  Maximal WS, with shoes - Cycle 1 | 0.02 (0.08)
  Maximal WS, with shoes - Cycle 2: number analyzed (Participants) | 286
  Maximal WS, with shoes - Cycle 2 | 0.03 (0.09)
  Maximal WS, with shoes - Cycle 3: number analyzed (Participants) | 217
  Maximal WS, with shoes - Cycle 3 | 0.03 (0.09)
  Maximal WS, with shoes - Cycle 4: number analyzed (Participants) | 134
  Maximal WS, with shoes - Cycle 4 | 0.04 (0.1)

27. Secondary Outcome: Mean Change From Baseline to Week 4 in Cadence
Description: All WS tests were conducted without walking aids over a distance of 10 metres at both a comfortable WS and at maximal WS. Evaluations of cadence were made barefoot and with shoes on, at baseline, at Weeks 4 and 12, at discretionary visits at Weeks 16, 20 and 24 of each cycle, and at EOS/EW. Outcome measure is reported per cycle as mean change from baseline at Week 4.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps/s
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
steps/s
  Comfortable WS, barefoot - Cycle 1: number analyzed (Participants) | 335
  Comfortable WS, barefoot - Cycle 1 | 0.08 (0.21)
  Comfortable WS, barefoot - Cycle 2: number analyzed (Participants) | 285
  Comfortable WS, barefoot - Cycle 2 | 0.08 (0.23)
  Comfortable WS, barefoot - Cycle 3: number analyzed (Participants) | 215
  Comfortable WS, barefoot - Cycle 3 | 0.08 (0.21)
  Comfortable WS, barefoot - Cycle 4: number analyzed (Participants) | 134
  Comfortable WS, barefoot - Cycle 4 | 0.07 (0.21)
  Comfortable WS, with shoes - Cycle 1: number analyzed (Participants) | 336
  Comfortable WS, with shoes - Cycle 1 | 0.07 (0.21)
  Comfortable WS, with shoes - Cycle 2: number analyzed (Participants) | 289
  Comfortable WS, with shoes - Cycle 2 | 0.08 (0.22)
  Comfortable WS, with shoes - Cycle 3: number analyzed (Participants) | 217
  Comfortable WS, with shoes - Cycle 3 | 0.08 (0.22)
  Comfortable WS, with shoes - Cycle 4: number analyzed (Participants) | 134
  Comfortable WS, with shoes - Cycle 4 | 0.07 (0.21)
  Maximal WS, barefoot - Cycle 1: number analyzed (Participants) | 336
  Maximal WS, barefoot - Cycle 1 | 0.07 (0.26)
  Maximal WS, barefoot - Cycle 2: number analyzed (Participants) | 286
  Maximal WS, barefoot - Cycle 2 | 0.08 (0.28)
  Maximal WS, barefoot - Cycle 3: number analyzed (Participants) | 215
  Maximal WS, barefoot - Cycle 3 | 0.09 (0.26)
  Maximal WS, barefoot - Cycle 4: number analyzed (Participants) | 134
  Maximal WS, barefoot - Cycle 4 | 0.11 (0.25)
  Maximal WS, with shoes - Cycle 1: number analyzed (Participants) | 335
  Maximal WS, with shoes - Cycle 1 | 0.07 (0.23)
  Maximal WS, with shoes - Cycle 2: number analyzed (Participants) | 286
  Maximal WS, with shoes - Cycle 2 | 0.09 (0.27)
  Maximal WS, with shoes - Cycle 3: number analyzed (Participants) | 217
  Maximal WS, with shoes - Cycle 3 | 0.09 (0.27)
  Maximal WS, with shoes - Cycle 4: number analyzed (Participants) | 134
  Maximal WS, with shoes - Cycle 4 | 0.09 (0.27)

28. Secondary Outcome: Mean Change From Baseline to Week 4 in Angle of Arrest (XV1), Angle of Catch (XV3) and Spasticity Angle (X) in the GSC (Knee Extended)
Description: Spasticity in the treated limb was assessed using the Tardieu Scale (TS) for the GSC (knee extended). The TS is administered by applying passive stretch to a muscle group at two velocities. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest, either due to subject discomfort or a mechanical resistance. The same movement is repeated at high velocity (as fast as possible) to determine the angle of catch and release. The angle of movement arrest at slow velocity (XV1) and the angle of catch at fast speed (XV3) were recorded at baseline, at Weeks 4 and 12 after each Dysport® injection, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. The spasticity angle (X) was calculated as the difference between XV1 and XV3. Mean changes in Angles XV1, XV3 and X from baseline to Week 4 are reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Degrees
  Angle of arrest (XV1) - Cycle 1: number analyzed (Participants) | 341
  Angle of arrest (XV1) - Cycle 1 | 2.7 (7.9)
  Angle of arrest (XV1) - Cycle 2: number analyzed (Participants) | 290
  Angle of arrest (XV1) - Cycle 2 | 2.4 (7.8)
  Angle of arrest (XV1) - Cycle 3: number analyzed (Participants) | 218
  Angle of arrest (XV1) - Cycle 3 | 2.6 (8.9)
  Angle of arrest (XV1) - Cycle 4: number analyzed (Participants) | 135
  Angle of arrest (XV1) - Cycle 4 | 2.7 (8.4)
  Angle of catch (XV3) - Cycle 1: number analyzed (Participants) | 341
  Angle of catch (XV3) - Cycle 1 | 7.1 (10.6)
  Angle of catch (XV3) - Cycle 2: number analyzed (Participants) | 289
  Angle of catch (XV3) - Cycle 2 | 7.3 (11.1)
  Angle of catch (XV3) - Cycle 3: number analyzed (Participants) | 218
  Angle of catch (XV3) - Cycle 3 | 7.9 (12.2)
  Angle of catch (XV3) - Cycle 4: number analyzed (Participants) | 135
  Angle of catch (XV3) - Cycle 4 | 9.5 (12.4)
  Spasticity angle (X) - Cycle 1: number analyzed (Participants) | 341
  Spasticity angle (X) - Cycle 1 | -4.4 (8.6)
  Spasticity angle (X) - Cycle 2: number analyzed (Participants) | 289
  Spasticity angle (X) - Cycle 2 | -4.9 (9.2)
  Spasticity angle (X) - Cycle 3: number analyzed (Participants) | 218
  Spasticity angle (X) - Cycle 3 | -5.4 (9.3)
  Spasticity angle (X) - Cycle 4: number analyzed (Participants) | 135
  Spasticity angle (X) - Cycle 4 | -6.8 (9.2)

29. Secondary Outcome: Mean Change From Baseline to Week 4 in Spasticity Grade (Y) in the GSC (Knee Extended)
Description: Spasticity in the treated limb was assessed using the TS for the GSC (knee extended). The TS is administered by applying passive stretch to a muscle group. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 =No resistance throughout passive movement, 1=slight resistance throughout passive movement, 2=clear catch at precise angle, interrupting passive movement, followed by release, 3=fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release. 4=unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. Spasticity grade (Y) was recorded at baseline, at Weeks 4 and 12 after each Dysport® injection, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. Mean changes in spasticity grade (Y) from baseline to Week 4 are reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Cycle 1: number analyzed (Participants) | 341
  Cycle 1 | -0.5 (0.8)
  Cycle 2: number analyzed (Participants) | 290
  Cycle 2 | -0.5 (0.7)
  Cycle 3: number analyzed (Participants) | 218
  Cycle 3 | -0.5 (0.7)
  Cycle 4: number analyzed (Participants) | 135
  Cycle 4 | -0.5 (0.8)

30. Secondary Outcome: Mean Change From Baseline to Week 4 in Angle of Arrest (XV1), Angle of Catch (XV3) and Spasticity Angle (X) in the Soleus Muscle (Knee Flexed)
Description: Spasticity in the treated limb was assessed using the TS for the soleus muscle (knee flexed). The TS is administered by applying passive stretch to a muscle group at two velocities. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest, either due to subject discomfort or a mechanical resistance. The same movement is repeated at high velocity (as fast as possible) to determine the angle of catch and release. The angle of movement arrest at slow velocity (XV1) and the angle of catch at fast speed (XV3) were recorded at baseline, at Weeks 4 and 12 after each Dysport® injection, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. The spasticity angle (X) was calculated as the difference between XV1 and XV3. Mean changes in Angles XV1, XV3 and X from baseline to Week 4 are reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Degrees
  Angle of arrest (XV1) - Cycle 1: number analyzed (Participants) | 341
  Angle of arrest (XV1) - Cycle 1 | 1.9 (8.0)
  Angle of arrest (XV1) - Cycle 2: number analyzed (Participants) | 290
  Angle of arrest (XV1) - Cycle 2 | 2.8 (8.1)
  Angle of arrest (XV1) - Cycle 3: number analyzed (Participants) | 218
  Angle of arrest (XV1) - Cycle 3 | 2.6 (8.5)
  Angle of arrest (XV1) - Cycle 4: number analyzed (Participants) | 135
  Angle of arrest (XV1) - Cycle 4 | 2.4 (8.6)
  Angle of catch (XV3) - Cycle 1: number analyzed (Participants) | 341
  Angle of catch (XV3) - Cycle 1 | 6.9 (10.3)
  Angle of catch (XV3) - Cycle 2: number analyzed (Participants) | 289
  Angle of catch (XV3) - Cycle 2 | 7.5 (10.8)
  Angle of catch (XV3) - Cycle 3: number analyzed (Participants) | 218
  Angle of catch (XV3) - Cycle 3 | 7.8 (11.2)
  Angle of catch (XV3) - Cycle 4: number analyzed (Participants) | 135
  Angle of catch (XV3) - Cycle 4 | 8.8 (11.4)
  Spasticity angle (X) - Cycle 1: number analyzed (Participants) | 341
  Spasticity angle (X) - Cycle 1 | -5.0 (10.0)
  Spasticity angle (X) - Cycle 2: number analyzed (Participants) | 289
  Spasticity angle (X) - Cycle 2 | -4.7 (9.8)
  Spasticity angle (X) - Cycle 3: number analyzed (Participants) | 218
  Spasticity angle (X) - Cycle 3 | -5.2 (9.6)
  Spasticity angle (X) - Cycle 4: number analyzed (Participants) | 135
  Spasticity angle (X) - Cycle 4 | -6.4 (11.1)

31. Secondary Outcome: Mean Change From Baseline to Week 4 in Spasticity Grade (Y) in the Soleus Muscle (Knee Flexed)
Description: Spasticity in the treated limb was assessed using the TS for the soleus muscle (knee flexed). The TS is administered by applying passive stretch to a muscle group. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 =No resistance throughout passive movement, 1=slight resistance throughout passive movement, 2=clear catch at precise angle, interrupting passive movement, followed by release, 3=fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release. 4=unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. Spasticity grade (Y) was recorded at baseline, at Weeks 4 and 12 after each Dysport® injection, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at EOS/EW. Mean changes in spasticity grade (Y) from baseline to Week 4 are reported per cycle.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
units on a scale
  Cycle 1: number analyzed (Participants) | 341
  Cycle 1 | -0.6 (0.8)
  Cycle 2: number analyzed (Participants) | 290
  Cycle 2 | -0.6 (0.7)
  Cycle 3: number analyzed (Participants) | 218
  Cycle 3 | -0.7 (0.8)
  Cycle 4: number analyzed (Participants) | 135
  Cycle 4 | -0.7 (0.7)

32. Secondary Outcome: Use of Walking Aids/Orthoses at Baseline and Week 4
Description: Subjects were assessed on their use of walking aids and orthoses at baseline, at Weeks 4 and 12 after each Dysport® injection, at discretionary visits at Weeks 16, 20 and 24 of each cycle and at the EOS/EW visit. Outcome measure is reported per cycle at baseline and Week 4. Number of subjects with no walking aid/orthoses were included in the 'No Walking Aid' category and number of subjects with any kind of walking aid/orthosis (including single point cane, tripod cane, ankle foot orthosis or other type of walking aid/orthosis) were combined into the 'Walking Aid' category.
Time Frame: Baseline and Week 4 of each cycle
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 345
Participants
  No Walking Aid at Baseline - Cycle 1 | 101
  Walking Aid at Baseline - Cycle 1 | 244
  No Walking Aid at Week 4 - Cycle 1: number analyzed (Participants) | 341
  No Walking Aid at Week 4 - Cycle 1 | 99
  Walking Aid at Week 4 - Cycle 1: number analyzed (Participants) | 341
  Walking Aid at Week 4 - Cycle 1 | 242
  No Walking Aid at Baseline - Cycle 2: number analyzed (Participants) | 297
  No Walking Aid at Baseline - Cycle 2 | 84
  Walking Aid at Baseline - Cycle 2: number analyzed (Participants) | 297
  Walking Aid at Baseline - Cycle 2 | 213
  No Walking Aid at Week 4 - Cycle 2: number analyzed (Participants) | 292
  No Walking Aid at Week 4 - Cycle 2 | 80
  Walking Aid at Week 4 - Cycle 2: number analyzed (Participants) | 292
  Walking Aid at Week 4 - Cycle 2 | 212
  No Walking Aid at Baseline - Cycle 3: number analyzed (Participants) | 224
  No Walking Aid at Baseline - Cycle 3 | 56
  Walking Aid at Baseline - Cycle 3: number analyzed (Participants) | 224
  Walking Aid at Baseline - Cycle 3 | 168
  No Walking Aid at Week 4 - Cycle 3: number analyzed (Participants) | 206
  No Walking Aid at Week 4 - Cycle 3 | 59
  Walking Aid at Week 4 - Cycle 3: number analyzed (Participants) | 206
  Walking Aid at Week 4 - Cycle 3 | 147
  No Walking Aid at Baseline - Cycle 4: number analyzed (Participants) | 139
  No Walking Aid at Baseline - Cycle 4 | 40
  Walking Aid at Baseline - Cycle 4: number analyzed (Participants) | 139
  Walking Aid at Baseline - Cycle 4 | 99
  No Walking Aid at Week 4 - Cycle 4: number analyzed (Participants) | 97
  No Walking Aid at Week 4 - Cycle 4 | 33
  Walking Aid at Week 4 - Cycle 4: number analyzed (Participants) | 97
  Walking Aid at Week 4 - Cycle 4 | 64

ADVERSE EVENTS:
Time Frame: From baseline to EOS (maximum duration of 52 weeks).
Description: AE data is reported as TEAEs. An AE was reported as a TEAE if it arose or the intensity increased during the treatment phase of this study.
Arm/Group | Total Dysport®
Serious Adverse Events (participants affected / at risk) | 43/345
Other Adverse Events (participants affected / at risk) | 69/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport® (N=345)
Venous thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Death
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 5 (5)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) — Death
Anxiety (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport® (N=345)
Fall (Injury, poisoning and procedural complications) | 42 (52)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 36 (41)

LIMITATIONS AND CAVEATS:
Data is summarised according to total dose received at each corresponding cycle (i.e. including 1000 U and 1500 U Dysport® in lower limb during all cycles, as well as 1000 U in lower limb + 500 U Dysport® in upper limb during Cycles 3 and 4).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No